CLINICAL TRIAL: NCT06687824
Title: Evaluation of the Effect of Black Tea Extract-Impregnated Gauze on Primary Bleeding Cessation After Molar Extraction: A Randomized Controlled Trial
Brief Title: Effect of Black Tea Extract Impregnated Gauze on Extracted Socket
Acronym: BTEIG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Manipal University College Malaysia (Other)
Responsible Party: Principal Investigator, Prof Dato' Dr. Rusdi Bin Abd. Raman, Professor Dato' Dr., Manipal University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MUCM/REC-042/2023
Record Dates: First submitted 2024-11-08; First posted 2024-11-14 (Actual); Results first posted 2025-05-20 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Extracted Socket
MeSH Terms: interventions — Tea

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Black Tea-Extract Impregnated Sterile Gauze (Experimental)
  Interventions: Other: Black Tea Extract
- 0.5% Povidone Iodine Impregnated Sterile Gauze (Placebo Comparator)
  Interventions: Other: 0.5% Povidone Iodine Impregnated Sterile Gauze

INTERVENTIONS:
Other: Black Tea Extract — Sterile gauze is impregnated into 5ml of black tea-extract solution with tannin concentration 18.67mg/ml
  Arms: Black Tea-Extract Impregnated Sterile Gauze
Other: 0.5% Povidone Iodine Impregnated Sterile Gauze — Diluted povidone-iodine act as negative control is added into sterile gauze to color blind the involved subject and the operator
  Arms: 0.5% Povidone Iodine Impregnated Sterile Gauze

SUMMARY:
Black tea is made from the leaves of a bush called Camellia sinensis. The main difference between green tea and black tea is that green tea is not completely oxidized while black tea is fully oxidized. Immediately after being harvested, the leaves of green tea are heated in order to halt the oxidation process, this ensures that the tea experiences minimal oxidation and stays a bright green color. Black tea, meanwhile, is allowed to fully oxidize after it is harvested. This means that the leaves turn brown or black, with green no longer present anywhere on the leaf. The chemical composition of black tea are tannins, theaflavins, carbohydrates, thearubigins, protein, flavonols, mineral matter, phenolic acids, volatiles, amino acids, methylxanthine. Among these, tannins play an important role in our research which helps in bleeding cessation after tooth extraction. Prolonged bleeding after tooth extraction can cause discomfort and thus affect patient's healthcare. Several methods have been proposed to enhance bleeding cessation, including the use of haemostatic agents and natural remedies such as tea. Black tea, in particular, has been suggested to have potential haemostatic properties due to its high content of tannins and flavonoids. However, the efficacy of black tea in promoting bleeding cessation after tooth extraction remains unclear. The purpose of this study is to evaluate the effect of black tea extract on primary bleeding cessation after extraction of molars. The study aims to investigate the potential benefits of black tea in reducing the bleeding time compared to a controlled group which uses normal sterile gauze. Our null hypothesis states that there is no difference in primary bleeding cessation time for black tea extract-impregnated sterile (BTE) gauze and 0.5% povidone iodine-impregnated sterile (PVI) gauze.

This study will be conducted in Oral Maxillofacial and Surgery Department in Polyclinic A, Faculty of Dentistry, Manipal University College Malaysia (MUCM). It involves forty-four randomly selected patients with molar extraction, satisfying the inclusion criteria and exclusion criteria stated. BTE gauze or PVI gauze will be placed at the freshly extracted socket after extraction. The state of bleeding of the socket is observed at 2,5 and 7 minutes.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or more
* ASA1 (American Society of Anesthesiologists physical status classification 1) and ASA2 patient

Exclusion Criteria:

* Sensitive to black tea
* Using complementary medical methods (herbal medicine, etc.) within the past month
* History of exposure of surgery site to radiation
* Using any antibiotic, corticosteroid, anticoagulant and contraceptive drug over the past month

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2024-04-02 (Actual); Primary Completion 2024-12-12 (Actual); Study Completion 2024-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sy Xuan Heng, Principal Investigator — Manipal University College Malaysia; Wan Ying Lim, Principal Investigator — Manipal University College Malaysia; Pei Wen Ho, Principal Investigator — Manipal University College Malaysia; Jia Xuan Lee, Principal Investigator — Manipal University College Malaysia; Cheryl Xue Rou Lee, Principal Investigator — Manipal University College Malaysia
Locations (1):
- Manipal University College Malaysia, Malacca, Malaysia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalalinia F, Amiri N, Mehrvarzian N, Fazly Bazzaz BS, Iranshahi M, Shahroodi A, Arabzadeh S, Abbaspour M, Badiee Aaval S, Movaffagh J. Topical green tea formulation with anti-hemorrhagic and antibacterial effects. Iran J Basic Med Sci. 2020 Aug;23(8):1085-1090. doi: 10.22038/ijbms.2020.41397.9782. PMID 32952956
- [Background] Kumbargere Nagraj S, Prashanti E, Aggarwal H, Lingappa A, Muthu MS, Kiran Kumar Krishanappa S, Hassan H. Interventions for treating post-extraction bleeding. Cochrane Database Syst Rev. 2018 Mar 4;3(3):CD011930. doi: 10.1002/14651858.CD011930.pub3. PMID 29502332
- [Background] Abbate R, Prisco D, Rostagno C, Boddi M, Gensini GF. Age-related changes in the hemostatic system. Int J Clin Lab Res. 1993;23(1):1-3. doi: 10.1007/BF02592271. PMID 8477086
- [Background] Le Blanc J, Lordkipanidze M. Platelet Function in Aging. Front Cardiovasc Med. 2019 Aug 7;6:109. doi: 10.3389/fcvm.2019.00109. eCollection 2019. PMID 31448291
- [Background] Chokotho L, van Hasselt E. The use of tannins in the local treatment of burn wounds - a pilot study. Malawi Med J. 2005 Jun;17(1):19-20. doi: 10.4314/mmj.v17i1.10866. PMID 27528993
- [Background] Marcinczyk N, Gromotowicz-Poplawska A, Tomczyk M, Chabielska E. Tannins as Hemostasis Modulators. Front Pharmacol. 2022 Jan 13;12:806891. doi: 10.3389/fphar.2021.806891. eCollection 2021. PMID 35095516
- [Background] Yerragudi N, Chawla JG, Kalidoss VK, Polineni S, Jayam C, Kumar C. The Optimal Hemostasis Duration After Tooth Extraction: A Randomized Controlled Trial. Cureus. 2023 Jan 3;15(1):e33331. doi: 10.7759/cureus.33331. eCollection 2023 Jan. PMID 36741661
- [Background] Chung KT, Wong TY, Wei CI, Huang YW, Lin Y. Tannins and human health: a review. Crit Rev Food Sci Nutr. 1998 Aug;38(6):421-64. doi: 10.1080/10408699891274273. PMID 9759559
- [Result] Soltani R, Haghighat A, Fanaei M, Asghari G. Evaluation of the effect of green tea extract on the prevention of gingival bleeding after posterior mandibular teeth extraction: a randomized controlled trial. Evid Based Complement Alternat Med. 2014;2014:857651. doi: 10.1155/2014/857651. Epub 2014 Jun 12. PMID 25024733
- [Result] Macpherson CR, Jacobs P. Bleeding time decreases with age. Arch Pathol Lab Med. 1987 Apr;111(4):328-9. PMID 3827541
- See also: Use of ultraviolet germicidal irradiation on disinfection — https://doi.org/10.1007/978-3-642-01999-9_1
- See also: Time Required for Haemostasis under Pressure from Dental Extraction Socket — http://doi.org/10.4103/ijdr.IJDR_93_18
- See also: Tannins may be employed medicinally in antidiarrheal, haemostatic, and antihemorrhoidal compounds — http://www.phytojournal.com/archives/2012/vol1issue3/PartA/8.1.pdf
- See also: 96 weeks of storage time when medical items are stored in clean, sterile storage medium — https://doi.org/10.1016/j.seta.2022.102924
- See also: Effect of green tea on second degree burn wound in rats — http://www.thieme-connect.com/products/ejournals/pdf/10.4103/0970-0358.146593.pdf
- See also: Quantitative estimation of tannins by HPLC — http://www.researchgate.net/publication/301544033_Quantitative_estimation_of_tannins_by_HPLC
- See also: in vivo study on the effect of African black tea extract on wound healing — http://www.medicalsciencejournal.com/archives/2020/vol6/issue6/6-4-52

RESULTS

PARTICIPANT FLOW:
Groups:
- 0.5% Povidone Iodine Impregnated Sterile Gauze: 5ml of 0.5% of povidone iodine solution is used for each gauze.
- Black Tea-Extract Impregnated Sterile Gauze: 5ml of black tea extract solution is used for each gauze with 18.67mg.ml tannin concentration.
Period: Overall Study
Arm/Group | 0.5% Povidone Iodine Impregnated Sterile Gauze | Black Tea-Extract Impregnated Sterile Gauze
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5% Povidone Iodine Impregnated Sterile Gauze | Black Tea-Extract Impregnated Sterile Gauze | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Customized [Count of Participants; unit: Participants]
  less than 21 years old | 1 | 5 | 6
  21-30 | 1 | 3 | 4
  31-40 | 2 | 3 | 5
  41-50 | 6 | 2 | 8
  51-60 | 6 | 4 | 10
  more than 60 years old | 6 | 5 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 18 | 29
  Male | 11 | 4 | 15
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Effect of Black Tea Extract-Impregnated Gauze on Primary Bleeding Cessation After Molar Extraction
Description: A stopwatch is used by the investigator to check the bleeding status of the extracted socket at 2, 5 and 7 minutes after compression of the socket with black tea extract-impregnated gauze or color-blinded sterile gauze
Time Frame: Primary bleeding cessation after extraction of molar is assessed up to 7 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% Povidone Iodine Impregnated Sterile Gauze | Black Tea-Extract Impregnated Sterile Gauze
Number analyzed (Participants) | 22 | 22
Participants
  less than 2 minutes | 17 | 12
  2-5 minutes | 4 | 10
  6-7 minutes | 1 | 0

2. Secondary Outcome: To Identify Adverse Effect of Black Tea-extract Impregnated Sterile Gauze and 0.5% Povidone Iodine Impregnated Sterile Gauze on Post-extraction Sites.
Description: Evaluate the presence of adverse effect 3 days after extraction via phone
Time Frame: 3 days post-extraction
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5% Povidone Iodine Impregnated Sterile Gauze | Black Tea-Extract Impregnated Sterile Gauze
Number analyzed (Participants) | 22 | 22
Participants
  Not present | 22 | 22
  present | 0 | 0

ADVERSE EVENTS:
Time Frame: 3 days post-extraction
Description: Participants were contacted via phone to evaluate the presence of adverse effect which was the presence of pain, irritation, burning sensation , itching sensation , fever and bad odor at the 3rd day after extraction.
Arm/Group | 0.5% Povidone Iodine Impregnated Sterile Gauze | Black Tea-Extract Impregnated Sterile Gauze
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-01): https://cdn.clinicaltrials.gov/large-docs/24/NCT06687824/Prot_SAP_000.pdf